CLINICAL TRIAL: NCT06071559
Title: Effects of Bariatric Surgery on obesity-and Diabetes-associated Abnormalities of Hemostasis, Inflammation and Vascular Function.
Brief Title: Bariatric Surgery on obesity-and Diabetes-associated Abnormalities of Hemostasis, Inflammation and Vascular Function.
Acronym: FIBRINO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ersta Diakoni (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anders Thorell, Consultant Surgeon, Clinical professor, Ersta Diakoni
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014/1793-31/1
Record Dates: First submitted 2023-04-13; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Surgery; Obesity Associated Disorder; Coagulation Disorder; Diabetes Complications
Keywords: Bariatric surgery; Fibrinolysis
MeSH Terms: conditions — Hemostatic Disorders; Diabetes Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obesitysurgery with diabetes (Other): One group with obesity and concomitant type 2 diabetes
  Interventions: Procedure: Laparoscopic Roux-en-y gastric bypass
- Obesitysurgery and non-diabetes (Other): One group with obesity alone
  Interventions: Procedure: Laparoscopic Roux-en-y gastric bypass

INTERVENTIONS:
Procedure: Laparoscopic Roux-en-y gastric bypass — Obesity surgery

SUMMARY:
The goal of this prospective cohort study is to examine circulating biomarkers before and after weight loss in patients with obesity, with or without concomitant diabetes, undergoing bariatric surgery. The main questions that are being addressed are:

* Do biomarkers of hemostasis, including coagulation, fibrinolysis, and platelet function improve following surgery and if so, is that improvement more pronounced in patients with diabetes?
* Do biomarkers of endothelial function and other aspects of vascular function improve following surgery and if so, is that improvement more pronounced in patients with diabetes?
* Do biomarkers of inflammation, including markers of adipocyte function, improve following surgery and if so, is that improvement more pronounced in patients with diabetes?
* The possible role of circulating extracellular vesicles reflecting biological functions above will also be investigated (optional) Participants will be asked to attend in total five study visits before and after surgery including a final visit at two years post-surgery. Comparisons will be performed within- as well as between groups.

DETAILED DESCRIPTION:
In this single centre, prospective, parallel group, cohort study, patients meeting the eligibility criteria are recruited at the department of surgery at Ersta hospital, Stockholm, Sweden. Patients with obesity and type 2 diabetes (T2D) are matched for age and sex with the group of patients with obesity without T2D. During the study the participants attend five study visits: at baseline, at the morning of surgery (after two weeks of low calory diet), 6 weeks, 1 year and 2 years after surgery. At each study visit a nurse records blood pressure, weight, height, and waist/hip circumferences. In addition, the nurse recalls the medical history and any medication use including contraceptive hormones and analgesics. Fat mass is determined using bioelectric impedance. Venous blood samples are collected with the patients in the supine position after overnight fasting and at least 20 minutes of rest. For later analyses, 25 mL of blood is collected in citrate tubes and centrifuged for 20 min at 2000 x g in room temperature. Plasma aliquots are subsequently stored at minus 80 degrees Celsius. Blood test regarding values at baseline (not the primary outcome variables) will be analysed at the local hospital laboratory. Examples of those basic variables are concentrations of glucose, insulin, blood cell counts and lipids.

ELIGIBILITY:
Inclusion criteria:

* Age 18-70 years old
* Planned for Roux-en-y gastric bypass surgery
* Obesity fulfilling criteria for bariatric surgery (according to the European Association for the Study of Obesity guidelines, ref. Yumuk et al. European Guidelines for Obesity Management in Adults. Obes Facts 2015;8:402-42.)

Exclusion criteria:

* Ongoing treatment with anticoagulant medication
* Ongoing treatment with antiplatelet medication other than acetylsalicylic acid
* Type 1 diabetes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Blood tests for endothelial function comparing two years after surgery with baseline (below referred to as "changes in"). | before surgery - 2 years after surgery
  Outcome measure:
  * Change in Hyaluronan (ng/ml)
  * Change in Syndacan-1 (ng/ml)
  * Change in E-selectin (ng/ml)
  * Change in Thrombomodulin (pg/ml)
  * Change in von Willebrand factor (%)
Blood tests for fibrinolysis comparing two years after surgery with baseline (below referred to as "changes in"). | before surgery - 2 years after surgery
  Outcome measure:
  * Change in PAI-1 activity (IU/ml)
  * Change in Fibrinogen (pg/ml)
  * Change in tPA activity (IU/ml)
  * Change in PAP complex (ng/ml)
  * Change in turbidimetric values - LagC (s)
  * Change in turbidimetric values - LagL (s)
  * Change in turbidimetric values - MaxAbsC (au)
  * Change in turbidimetric values - MaxAbsL (au
  * Change in turbidimetric values - Lys50MA (s)
  * Change in turbidimetric values - CRC (au/s)
  * Change in turbidimetric values - CRL (au/s)
Blood tests for inflammation comparing two years after surgery with baseline (below referred to as "changes in"). | before surgery - 2 years after surgery
  Outcome measure:
  * Change in high sensitivity CRP (microg/ml)
  * Change in soluble IL6 receptor (ng/mL)
  * Change in IL6 (pg/mL)
  * Change in soluble gp130 (ng/mL)
  * Change in TNFalfa (pg/ml)
Blood tests for extracellular vesicles comparing two years after surgery with baseline (below referred to as "changes in"). | before surgery - 2 years after surgery
  Exploratory analyses of extracellular vesicles (EV) in plasma using flow cytometry. EV exposing antigens of cell specific origin and/or biologically active molecules will be assessed. Outcome measure: Change in number of EVs (number of EV/micoL)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Thorell, Professor, Principal Investigator — Karolinska Institutet Danderyds sjukhus/Ersta sjukhus

IPD SHARING:
Plan to Share IPD: No